CLINICAL TRIAL: NCT03097380
Title: An Open-label Positron Emission Tomography Phase I Study to Determine Muscarinic Receptor Occupancy in the Lungs in Healthy Volunteers After Inhalation of Single Dose of Tiotropium or AZD2115.
Brief Title: PET Study to Determine Muscarinic Receptor Occupancy in Lungs After Inhalation of AZD2115 and Tiotropium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3060C00014
Record Dates: First submitted 2017-03-06; First posted 2017-03-31 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer study
MeSH Terms: interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZD2115 (Experimental)
  Interventions: Drug: AZD2115; Radiation: [11C]AZ13754366
- Spiriva (Tiotropium) (Active Comparator)
  Interventions: Drug: SPIRIVA; Radiation: [11C]AZ13754366
- [11C]AZ13754366 (Experimental)
  Interventions: Radiation: [11C]AZ13754366

INTERVENTIONS:
Drug: AZD2115 — AZD2115
  Arms: AZD2115
Drug: SPIRIVA — Tiotropium
  Arms: Spiriva (Tiotropium)
Radiation: [11C]AZ13754366 — Radioligand

SUMMARY:
An open-label study using positionemissiontomography (PET) to explore the binding of AZD2115 and Tiotropium to muscarinic receptors in the lungs in healthy volunteers after inhalation.

DETAILED DESCRIPTION:
A phase I open-label exploratory study in healthy male volunteers using positionemissiontomography (PET). The study will test the hypothesis that Tiotropium and AZD2115 binds to the mAchRs in a saturable manner and aims to examine the relationship between receptor occupancy and drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures
* Healthy male subjects, aged 20 to 50 years (inclusive)
* Male subjects must be surgically sterile or use an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the first dose) and for 3 months after the last dose of study drug to prevent pregnancy in a partner
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50.0 kg and no more than 100.0 kg, inclusive
* Able and willing to participate in all scheduled evaluations and abide by all study restrictions
* Ability to inhale from the study drug training devices at visit 1
* Subjects who are blood donors should not donate blood during the study and for 3 months following their last dose of study drug.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the study results or the subject's ability to participate in the study.
* Any clinical significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP)
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator.
* Any positive results on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV)
* Abnormal vital signs, after 10 minutes of supine rest, defined as any of the following:

  * Systolic blood pressure (BP) <90 mmHg or >140 mmHg
  * Diastolic BP <50 mmHg or >90 mmHg
  * Heart rate <45 bpm or > 100 bpm
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes, as determined by the investigator. This may include subjects with any of the following:

  * PR (PQ) interval prolongation of clinical significance as judged by the Investigator
  * Intermittent second or third degree AV block (AV block II Mobitz type 1 Wenchebach, while asleep or in deep rest is not disqualifying)
  * Incomplete, full, or intermittent bundle branch block (QRS less than 110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy)
  * Abnormal T wave morphology, particularly in the protocol-defined primary lead
  * Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) greater than 450 ms or shortened QTcF less than 340 ms or a family history of long QT syndrome.
* History of alcohol abuse or excessive intake of alcohol, as judged by the investigator.
* Positive screen for drugs of abuse at visit 1.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, other than seasonal allergies, as judged by the Investigator, or history of hypersensitivity to drugs with similar chemical structure or class as AZD2115.
* Use of any prescribed or non-prescribed medication, during the 4 weeks (or longer depending on the medication's half-life) prior to the administration of IMP.
* Use of drugs with enzyme inducing properties such as St John's Wort within 4 weeks prior to the investigational product administration.
* Current smokers or subjects who have smoked or used nicotine products within 6 months prior to visit 1
* Plasma donation within 1 month of screening or any blood donation/blood loss equal to or greater than 500 mL during the 3 months prior to screening.
* Previous enrolment in the present study
* Involvement in the planning and/or conduct of the study
* Participation in another clinical study with an investigational product during the last 3 months
* Negative Allen test in both hands
* Claustrophobia that would contraindicate PET measurement.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Reduction in distribution volume (VT)% | up to 9 h post dose
  To describe the AZD2115 dose-muscarinic receptor occupancy relationship in the lungs in healthy volunteers

SECONDARY OUTCOMES:
Receptor occupancy (RO) % | up to 9 h post dose
  To describe the muscarinic receptor occupancy after inhalation of AZD2115 and Tiotropium in the lungs in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cselenyi Z, Jucaite A, Ewing P, Stenkrona P, Kristensson C, Johnstrom P, Schou M, Bolin M, Halldin C, Larsson B, Grime K, Eriksson UG, Farde L. Proof of lung muscarinic receptor occupancy by tiotropium: Translational Positron Emission Tomography studies in non-human primates and humans. Front Nucl Med. 2023 Jan 18;2:1080005. doi: 10.3389/fnume.2022.1080005. eCollection 2022. PMID 39354985
- [Derived] Cselenyi Z, Jucaite A, Kristensson C, Stenkrona P, Ewing P, Varrone A, Johnstrom P, Schou M, Vazquez-Romero A, Moein MM, Bolin M, Siikanen J, Gryback P, Larsson B, Halldin C, Grime K, Eriksson UG, Farde L. Quantification and reliability of [11C]VC - 002 binding to muscarinic acetylcholine receptors in the human lung - a test-retest PET study in control subjects. EJNMMI Res. 2020 Jun 3;10(1):59. doi: 10.1186/s13550-020-00634-0. PMID 32495011